CLINICAL TRIAL: NCT06130566
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, 3-arm, Multinational, Multicenter Study to Evaluate the Efficacy and Safety of Amlitelimab Monotherapy by Subcutaneous Injection in Participants Aged 12 Years and Older With Moderate-to-severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Efficacy and Safety of Subcutaneous Amlitelimab Monotherapy Compared With Placebo in Participants Aged 12 Years and Older With Moderate-to-severe Atopic Dermatitis
Acronym: COAST 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17559; U1111-1275-9715 (Registry Identifier: ICTRP); 2022-501196-41 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Amlitelimab dose 1 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab
- Amlitelimab dose 2 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab
- Placebo (Placebo Comparator): Subcutaneous injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlitelimab — Injection solution SC injection
  Other Names: SAR445229
  Arms: Amlitelimab dose 1; Amlitelimab dose 2
Drug: Placebo — Injection solution SC injection
  Arms: Placebo

SUMMARY:
This is a parallel group, Phase 3, multinational, multicenter, randomized, double blind, placebo-controlled, 3-arm monotherapy study for treatment of participants diagnosed with moderate to severe atopic dermatitis (AD), whose disease is not adequately controlled with topical prescription therapies or when those therapies are not advisable.

The purpose of this study is to measure the efficacy and safety of treatment with amlitelimab solution for SC injection compared with placebo in participants with moderate to severe AD aged 12 years and older.

Study details include:

At the end of the treatment period, participants will have an option to enter a separate study: the blinded extension study EFC17600 (ESTUARY).

For participants not entering the blinded extension Study EFC17600 (ESTUARY), the study duration will be up to 44 weeks including a 2 to 4-week screening, a 24-week randomized double-blind period, and a 16-week safety follow-up.

For participants entering the blinded extension Study EFC17600 (ESTUARY), the study duration will be up to 28 weeks including a 2 to 4-week screening and a 24-week randomized double-blind period.

The total treatment duration will be up to 24 weeks. The total number of visits will be up to 10 visits (or 9 visits for those entering the blinded extension study EFC17600] (ESTUARY).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 12 years of age (when signing informed consent form)
* Diagnosis of AD for at least 1 year (defined by the American Academy of Dermatology Consensus Criteria)
* Documented history (within 6 months before screening) of either inadequate response or inadvisability to topical treatments, and/or inadequate response to systemic therapies (within 12 months before screening)
* v-IGA-AD of 3 or 4 at baseline visit
* EASI score of 16 or higher at baseline
* AD involvement of 10% or more of BSA at baseline
* Weekly average of daily PP-NRS of ≥ 4 at baseline visit.
* Able and willing to comply with requested study visits and procedures
* Body weight ≥25 kg

Exclusion Criteria:

* Skin co-morbidity that would adversely affect the ability to undertake AD assessments
* Known history of or suspected significant current immunosuppression
* Any malignancies or history of malignancies prior to baseline (with the exception of non-melanoma skin cancer excised and cured >5 years prior to baseline)
* History of solid organ or stem cell transplant
* Any active or chronic infection including helminthic infection requiring systemic treatment within 4 weeks prior to baseline (1 week in the event of superficial skin infections)
* Positive for human immunodeficiency virus (HIV), Hepatitis B or hepatitis C at screening visit
* Having active tuberculosis (TB), latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection, or who are at high risk of contracting TB
* Having received any of the specified therapy within the specified timeframe(s) prior to the baseline visit
* In the Investigator's opinion, any clinically significant laboratory results or protocol specified laboratory abnormalities at screening
* History of hypersensitivity or allergy to any of the excipients or investigational medicinal product (IMP)

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
EU, EU reference countries, and Japan: Proportion of participants with Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points at Week 24 | Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
EU, EU reference countries, and Japan: Proportion of participants reaching 75% reduction from baseline in Eczema Area and Severity Index (EASI) score (EASI-75) at Week 24 | Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
US and US reference countries: Proportion of participants with vIGA-AD of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points at Week 24 | Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).

SECONDARY OUTCOMES:
Proportion of participants reaching EASI-75 at Week 24 (for US and US reference countries only) | Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score.
Proportion of participants with vIGA-AD 0 (clear) or 1 (almost clear) with presence of only barely perceptible erythema (no induration/papulation, no lichenification, no oozing or crusting) and a reduction from baseline of ≥2 points | Baseline to Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants with ≥4-point reduction in weekly average of daily Peak Pruritus-Numerical Rating Scale (PP-NRS) from baseline in participants with baseline weekly average of daily PP-NRS ≥4 | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Proportion of participants reaching EASI-75 | Baseline to Week 20
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score.
Proportion of participants with vIGA-AD of 0 (clear) or 1 (almost clear) and a reduction from baseline of ≥2 points | Baseline to Week 20
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants reaching EASI-90 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-90 is 90% reduction from baseline in EASI score.
Proportion of participants reaching EASI-100 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-100 is 100% reduction from baseline in EASI score.
Proportion of participants with PP-NRS 0 or 1 | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Change in Dermatology Life Quality Index (DLQI) from baseline in participants with age ≥16 years old | Baseline to Week 24
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Proportion of participants with a reduction in DLQI ≥4 from baseline in participants with age ≥16 years old and with DLQI baseline ≥4 | Baseline to Week 24
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Change in Children Dermatology Life Quality Index (CDLQI) from baseline in participants with age ≥12 to <16 years old | Baseline to Week 24
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in children aged 4-<16 years. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Proportion of participants with a reduction in CDLQI ≥6 from baseline in participants with age ≥12 to <16 years old and with CDLQI baseline ≥6 | Baseline to Week 24
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in children aged 4-<16 years. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Change in Hospital Anxiety Depression Scale (HADS) from baseline | Baseline to Week 24
  The HADS is 14-item questionnaire with two subscales: anxiety & depression. Each subscale (anxiety & depression) ranges 0-21. The total HADS score ranges 0-42 with higher score indicating a poorer state.
Proportion of participants with HADS subscale Anxiety (HADS-A) <8 in participants with baseline HADS-A ≥8 | Baseline to Week 24
  HADS-A score ranges 0-21 with higher score indicating a poorer state.
Proportion of participants with HADS subscale Depression (HADS-D) <8 in participants with HADS-D baseline ≥8 | Baseline to Week 24
  HADS-D score ranges 0-21 with higher score indicating a poorer state.
Absolute change in weekly average of daily Skin Pain-Numerical Rating Scale (SP-NRS) from baseline | Baseline to Week 24
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Proportion of participants with a reduction in weekly average of daily SP-NRS ≥4 from baseline in participants with baseline weekly average of daily SP-NRS ≥4 | Baseline to Week 24
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Percent change in weekly average of daily SP-NRS from baseline | Baseline to Week 24
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Proportion of participants with vIGA-AD 0 | Week 24
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Absolute change in weekly average of daily Sleep Disturbance-Numerical Rating Scale (SD-NRS) from baseline | Baseline to Week 24
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Proportion of participants with a reduction in weekly average of daily SD-NRS ≥3 from baseline in participants with Baseline weekly average of daily SD-NRS ≥3 | Baseline to Week 24
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Percent change in weekly average of daily SD-NRS | Baseline to Week 24
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Percent change in EASI score from baseline | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Percent change in weekly average of daily PP-NRS from baseline | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Absolute change in weekly average of daily PP-NRS from baseline | Baseline to Week 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Proportion of participants reaching EASI-50 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-50 is 50% reduction from baseline in EASI score.
Proportion of participants with EASI ≤7 | Baseline to Week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Change in percent Body Surface Area (BSA) affected by AD from baseline | Baseline to Week 24
Percent change in Scoring Atopic Dermatitis (SCORAD) index from baseline | Baseline to Week 24
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Absolute change in SCORAD index from baseline | Baseline to Week 24
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Proportion of participants with a reduction in SCORAD ≥ 8.7 points from baseline in participants with baseline SCORAD score ≥ 8.7 | Baseline to Week 24
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Change in Patient Oriented Eczema Measure (POEM) from baseline | Baseline to Week 24
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Proportion of participants with a reduction in POEM ≥4 from baseline in participants with POEM Baseline ≥4 | Baseline to Week 24
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Proportion of participants with rescue medication use | Baseline to Week 24
Percentage of participants who experienced Treatment-Emergent Adverse Events (TEAEs), experienced Treatment-Emergent Serious Adverse Events (TESAEs) and/or Treatment-Emergent Adverse Events of Special Interest (AESI) | Baseline to Week 40
Serum amlitelimab concentrations | Baseline to Week 40
Incidence of antidrug antibodies (ADAs) of amlitelimab | Baseline to Week 40

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (148):
- United States (42):
  - Scottsdale Clinical Trials- Site Number : 8401149, Scottsdale, Arizona
  - First OC Dermatology- Site Number : 8401025, Fountain Valley, California
  - Center for Dermatology Clinical Research- Site Number : 8401018, Fremont, California
  - Sunwise Clinical Research- Site Number : 8401022, Lafayette, California
  - Carbon Health - North Hollywood - NoHo West- Site Number : 8401218, North Hollywood, California
  - Northridge Clinical Trials - Northridge- Site Number : 8401080, Northridge, California
  - St Jude Clinical Research- Site Number : 8401287, Doral, Florida
  - Beth Israel Deaconess Medical Center - Fort Myers- Site Number : 8401286, Fort Myers, Florida
  - Direct Helpers Research Center- Site Number : 8401056, Hialeah, Florida
  - Encore Medical Research- Site Number : 8401030, Hollywood, Florida
  - Florida International Research Center- Site Number : 8401091, Miami, Florida
  - Miami Dermatology and Laser Research- Site Number : 8401086, Miami, Florida
  - Clinical Neuroscience Solutions - Orlando - South Delaney Avenue- Site Number : 8401035, Orlando, Florida
  - Cleaver Medical Group Dermatology- Site Number : 8401139, Cumming, Georgia
  - Skin Care Physicians of Georgia - Macon- Site Number : 8401034, Macon, Georgia
  - Javara Research - Thomasville- Site Number : 8401189, Thomasville, Georgia
  - Rophe Adult & Pediatric Medicine- Site Number : 8401289, Union City, Georgia
  - Skin Sciences- Site Number : 8401039, Louisville, Kentucky
  - MedPharmics - Covington- Site Number : 8401137, Covington, Louisiana
  - MedPharmics - Lafeyette- Site Number : 8401152, Lafayette, Louisiana
  - Massachusetts General Hospital- Site Number : 8401192, Boston, Massachusetts
  - Metro Boston Clinical Partners- Site Number : 8401128, Needham, Massachusetts
  - Revival Research - Doral- Site Number : 8401012, Dearborn, Michigan
  - Henry Ford Hospital- Site Number : 8401044, Detroit, Michigan
  - SKY Integrative Medical Center/SKYCRNG - Ridgeland- Site Number : 8401058, Ridgeland, Mississippi
  - MediSearch Clinical Trials- Site Number : 8401140, Saint Joseph, Missouri
  - Somnos Clinical Research- Site Number : 8401203, Lincoln, Nebraska
  - Universal Dermatology- Site Number : 8401224, Fairport, New York
  - Sadick Research Group - New York - Park Avenue- Site Number : 8401050, New York, New York
  - CHEAR Center- Site Number : 8401123, The Bronx, New York
  - Onsite Clinical Solutions - Charlotte - Blakeney Park Drive- Site Number : 8401124, Charlotte, North Carolina
  - Oregon Medical Research Center- Site Number : 8401017, Portland, Oregon
  - Vial Health - DermDox Dermatology- Site Number : 8401031, Camp Hill, Pennsylvania
  - Paddington Testing Company- Site Number : 8401041, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia- Site Number : 8401193, Philadelphia, Pennsylvania
  - Tribe Clinical Research - 525 Verdae Boulevard- Site Number : 8401225, Greenville, South Carolina
  - Dermatology Treatment and Research Center- Site Number : 8401164, Dallas, Texas
  - Skin Specialist of Addison- Site Number : 8401208, Dallas, Texas
  - Texas Dermatology and Laser Specialists- Site Number : 8401131, San Antonio, Texas
  - Stryde Research - Epiphany Dermatology- Site Number : 8401185, Southlake, Texas
  - Springville Dermatology - Springville- Site Number : 8401106, Springville, Utah
  - Virginia Dermatology & Skin Cancer Center- Site Number : 8401047, Norfolk, Virginia
- Argentina (4):
  - Investigational Site Number : 0320023, Buenos Aires, Buenos Aires F.D.
  - Investigational Site Number : 0320024, SAN Miguel de Tucumã¡n, Tucumán Province
  - Investigational Site Number : 0320022, Buenos Aires
  - Investigational Site Number : 0320010, Buenos Aires
- Australia (5):
  - Investigational Site Number : 0360010, Westmead, New South Wales
  - Investigational Site Number : 0360007, Woolloongabba, Queensland
  - Investigational Site Number : 0360008, Melbourne, Victoria
  - Investigational Site Number : 0360006, Melbourne, Victoria
  - Investigational Site Number : 0361006, Traralgon, Victoria
- Brazil (10):
  - Centro de Pesquisas da Clínica IBIS- Site Number : 0760002, Salvador, Estado de Bahia
  - Hospital São Domingos- Site Number : 0760028, Bequimão, Maranhão
  - Hospital de Clinicas da Universidade Federal do Parana- Site Number : 0760022, Curitiba, Paraná
  - PUC Trials- Nucleo de Pesquisa clinica da Escola de Medicina da PUCPR- Site Number : 0760023, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre- Site Number : 0760005, Porto Alegre, Rio Grande do Sul
  - Clinica de Alergia Martti Antila- Site Number : 0760006, Sorocaba, São Paulo
  - CCBR / IBPClin - Instituto Brasil de Pesquisa Clínica- Site Number : 0760018, Rio de Janeiro
  - Faculdade de Medicina do ABC- Site Number : 0760001, Santo André
  - Centro de Desenvolvimento em Estudos ClÌnicos Brasil- Site Number : 0760014, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo- Site Number : 0760012, São Paulo
- Canada (12):
  - Investigational Site Number : 1240031, Edmonton, Alberta
  - Investigational Site Number : 1240040, Surrey, British Columbia
  - Investigational Site Number : 1240033, Ajax, Ontario
  - Investigational Site Number : 1240055, Hamilton, Ontario
  - Investigational Site Number : 1240029, London, Ontario
  - Investigational Site Number : 1241108, Niagara Falls, Ontario
  - Investigational Site Number : 1240034, Ottawa, Ontario
  - Investigational Site Number : 1240013, Toronto, Ontario
  - Investigational Site Number : 1240035, Toronto, Ontario
  - Investigational Site Number : 1240043, Saint-Jérôme, Quebec
  - Investigational Site Number : 1240028, Regina, Saskatchewan
  - Investigational Site Number : 1240036, Saskatoon, Saskatchewan
- Chile (10):
  - Investigational Site Number : 1520009, Osorno, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520010, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520011, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520012, Talcahuano
- China (8):
  - Investigational Site Number : 1560042, Beijing
  - Investigational Site Number : 1560060, Chengdu
  - Investigational Site Number : 1560068, Chengdu
  - Investigational Site Number : 1560057, Chongqing
  - Investigational Site Number : 1560065, Chongqing
  - Investigational Site Number : 1560058, Guangzhou
  - Investigational Site Number : 1560059, Jinan
  - Investigational Site Number : 1560064, Shenzhen
- France (5):
  - Investigational Site Number : 2500008, Antony
  - Investigational Site Number : 2500009, Nantes
  - Investigational Site Number : 2500003, Paris
  - Investigational Site Number : 2500007, Reims
  - Investigational Site Number : 2500010, Romans-sur-Isère
- Germany (7):
  - Investigational Site Number : 2760009, Bad Bentheim
  - Investigational Site Number : 2760014, Buxtehude
  - Investigational Site Number : 2760017, Hamburg
  - Investigational Site Number : 2762208, Kiel
  - Investigational Site Number : 2760018, Magdeburg
  - Investigational Site Number : 2760016, Mainz
  - Investigational Site Number : 2762201, Münster
- Greece (4):
  - Investigational Site Number : 3000004, Athens
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000002, Thessaloniki
  - Investigational Site Number : 3000003, Thessaloniki
- India (8):
  - Investigational Site Number : 3560001, Ahmedabad
  - Investigational Site Number : 3560005, Belagavi
  - Investigational Site Number : 3560008, Bengaluru
  - Investigational Site Number : 3560004, Chandigarh
  - Investigational Site Number : 3560006, Haryāna
  - Investigational Site Number : 3560007, Kolkata
  - Investigational Site Number : 3560002, Nagpur
  - Investigational Site Number : 3560003, Pune
- Israel (6):
  - Investigational Site Number : 3760004, Afula
  - Investigational Site Number : 3760005, Beersheba
  - Investigational Site Number : 3760001, Haifa
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760006, Petah Tikva
  - Investigational Site Number : 3760002, Petah Tikva
- Poland (9):
  - Investigational Site Number : 6160006, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160003, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6162406, Krakow
  - Investigational Site Number : 6160002, Lodz
  - Investigational Site Number : 6160004, Lublin
  - Investigational Site Number : 6160011, Olsztyn
  - Investigational Site Number : 6160010, Tarnów
  - Investigational Site Number : 6160009, Warsaw
  - Investigational Site Number : 6160007, Warsaw
- South Korea (13):
  - Investigational Site Number : 4100008, Daegu, Daegu
  - Investigational Site Number : 4100002, Ansan-si, Gyeonggi-do
  - Investigational Site Number : 4100014, Seongnam-si, Gyeonggi-do
  - Investigational Site Number : 4100009, Suwon, Gyeonggi-do
  - Investigational Site Number : 4100003, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 4100015, Bupyeong-gu, Incheon-gwangyeoksi
  - Investigational Site Number : 4100010, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100013, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100007, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100011, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100017, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100012, Gwangju
- Taiwan (5):
  - Investigational Site Number : 1583201, Kaohsiung City
  - Investigational Site Number : 1583202, Taichung
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580003, Taipei
  - Investigational Site Number : 1583203, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17559 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25523&tenant=MT_SNY_9011